CLINICAL TRIAL: NCT01655784
Title: Framing Eighteen Coils in Cerebral Aneurysms Trial: FEAT
Brief Title: Framing Eighteen Coils in Cerebral Aneurysms Trial
Acronym: FEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Stryker Neurovascular (Industry)
Responsible Party: Principal Investigator, JD Mocco, Associate Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 120439
Record Dates: First submitted 2012-07-20; First posted 2012-08-02 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Cerebral Aneurysm
Keywords: aneurysm; intracranial aneurysm; cerebral aneurysm; intracranial embolization; aneurysm embolization; intracranial coil; eighteen coils; bare platinum coils; GDC Coil; Target Coil
MeSH Terms: conditions — Intracranial Aneurysm; Aneurysm

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Eighteen Coils (0.014-0.0155 inch) (Active Comparator): Subjects who randomize to this arm will receive larger diameter bare platinum coils for treatment of their cerebral aneurysm. Subjects in this arm could receive a combination of the following protocol approved intracranial coils depending on the phase: Target XL 360 Standard, Target XL 360 Soft, Target XL 360 Helical, GDC-18 360 Standard, GDC-18 3D, GDC-18 2D, GDC-18 Soft, and/or 0.014-0.0155 inch diameter bare platinum intracranial coils.
  Interventions: Procedure: Coil Embolization with larger Diameter Coils
- Standard Coils (0.014 inch) (Active Comparator): Subjects who randomize to this arm will receive the standard diameter bare platinum coils for treatment of their cerebral aneurysm. Subjects in this arm could receive a combination of the following protocol approved intracranial coils depending on the phase: Target 360 Standard, Target 360 Soft, Target 360 Ultra, Target 360 NANO, Target 360 Helical Ultra, GDC-10 360 Standard SR, GDC-10 360 Soft SR, GDC-10 UltraSoft, GDC-10 3D, GDC-10 2D, GDC-10 Soft 2D SR, GDC-10 Soft SR, GDC-10 Soft, and/or any additional 0.014 inch or less diameter bare platinum intracranial coils.
  Interventions: Procedure: Coil Embolization with Standard Diameter Coils

INTERVENTIONS:
Procedure: Coil Embolization with larger Diameter Coils — Eighteen Coils placed in cerebral aneurysm
  Other Names: Eighteen Coils; Cerebral Aneurysm Embolization; Aneurysm Coils
  Arms: Eighteen Coils (0.014-0.0155 inch)
Procedure: Coil Embolization with Standard Diameter Coils — Cerebral aneurysms will be embolized with standard diameter coils.
  Other Names: Eighteen Coils; Cerebral Aneurysm Embolization; Aneurysm Coils
  Arms: Standard Coils (0.014 inch)

SUMMARY:
This trial is being conducted in order to compare angiographic outcomes in patients receiving 0.014-0.0155" platinum framing and filling coils (larger diameter coils) versus those treated solely with coils less than 0.014" (with a standard diameter).

Hypothesis: Angiographic occlusion at follow-up imaging will be more frequent in patients receiving 0.014-0.0155" platinum coils during embolization compared to those receiving smaller-diameter coils.

DETAILED DESCRIPTION:
Primary Study Objective: Occlusion rate: angiographic occlusion, improvement or no change in the post-coiling appearance of the aneurysm as judged by an independent core lab on follow-up angiography at 12-18 months after endovascular embolization.

Secondary Objectives:

1. Treatment related morbidity and mortality, as measured by the NIH stroke scale.
2. Packing density as measured by volumetric filling of the aneurysm.
3. Clinical outcome at 3-6 and 12-18 months post-coiling, as measured by the modified Rankin scale.
4. Re-hemorrhage and re-treatment rates.

Study Design: FEAT will be a prospective, randomized trial comparing the utilization of 0.014-0.0155" coils versus smaller diameter coils in mid-sized aneurysm treatment. The 0.014-0.0155" bare platinum coils (Stryker, Natick, MA) are FDA-approved and in common use at institutions in this country and across the world. Patients will be enrolled who meet the inclusion criteria and consent to participate. Patients will be randomly assigned by a central web-based system in a 1:1 manner to either the framing coil treatment or the non-framing coil treatment. Data on each patient will be collected at the time of enrollment and treatment, and at first and second follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Patient presenting with ruptured or unruptured cerebral aneurysm appropriate for endovascular treatment as determined by the neurovascular treating team (neurointerventionist and/or neurosurgeon).
2. The neurointerventionist feels that the aneurysm can be safely treated with either using, or not using, a 0.015-0.0155" platinum coil.
3. Patients are 18-80 years of age (inclusive).
4. Patient must be Hunt and Hess grade 0 to 3.
5. Patient has given fully informed consent to endovascular coiling procedure. If the patient cannot consent for themselves, appropriate written consent has been sought from their next of kin or appropriate power of attorney.
6. Aneurysm 6-14 mm in maximum diameter.
7. Patient is willing and able to return for clinical evaluation and follow-up imaging evaluation (angiography or MRA) at 3-6 months and 12-18 months after endovascular treatment.
8. The patient has not been previously randomized into this trial or another related ongoing trial.
9. The aneurysm has not been previously treated by coiling or clipping.

Exclusion Criteria:

1. Patient has more than one aneurysm requiring treatment in the current treatment session, and only one of those to be treated aneurysms fits the FEAT inclusion criteria (ie - if either (1) a patient has multiple aneurysms, but only one will be treated at enrollment; or (2) if two or more aneurysms are treated during the current treatment session and BOTH are able to be enrolled, then they remain eligible for the trial). Non-treated additional aneurysms may be treated at a later date with any coil type that the operator chooses).
2. Target aneurysm has had previous coil treatment or has been surgically clipped.
3. Hunt and Hess score is 4 or 5 after subarachnoid hemorrhage.
4. Inability to obtain informed consent.
5. Medical or surgical co-morbidity such that the patient's life expectancy is less than 2 years.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 651 (Actual)
Dates: Start 2012-12-04 (Actual); Primary Completion 2024-02-19 (Actual); Study Completion 2024-02-19 (Actual)

PRIMARY OUTCOMES:
Occlusion Rate | 12-18 Month Follow-up
  Occlusion rate: Angiographic occlusion, improvement or no change in the post-coiling appearance of the aneurysm as judged by an independent core lab on follow-up angiography at 12-18 months after endovascular embolization.

SECONDARY OUTCOMES:
Morbidity | Entire Study Duration (from signed research consent until 12-18 month follow-up complete)
  Morbidity will be measured by the NIH Stroke Scale and tracked regardless of whether it is related to the study procedure.
Packing Density | Post-Procedure (images taken during the procedure immediately after the coils are placed will be assessed)
  Packing density will be measured by volumetric filling of the aneurysm by reviewing post-op angiographic films.
Clinical Outcome | 3-6 Month Follow-up and 12-18 Month Follow-up
  Clinical outcome at both follow-up time points will be measured by the modified Rankin Scale.
Re-hemorrhage and Re-treatment Rates | 3-6 Month Follow-up and 12-18 Month Follow-up
  Re-hemorrhage rates will be tracked and recorded during both follow-up time points.
Mortality | Entire Study Duration (from study procedure until 12-18 month follow-up)
  Mortality will be tracked throughout the study and recorded regardless of whether it is related to treatment.
Retreatment | 3-6 Month Follow-up and 12-18 Month Follow-up
  Retreatment rates will be tracked and recorded during both follow-up time points.

CONTACTS AND LOCATIONS:
Overall Officials: J D Mocco, MD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (24):
- United States (24):
  - UCSF-Fresno, Community Regional Medical Center, Fresno, California
  - Radiology Imaging Associates, Englewood, Colorado
  - Colorado Neurological Institute, Englewood, Colorado
  - University of Florida, Gainesville, Florida
  - University of South Florida - Tampa General, Tampa, Florida
  - University of Kentucky, Lexington, Kentucky
  - University of Massachusetts Medical School, North Worcester, Massachusetts
  - University of Mississippi, Jackson, Mississippi
  - University of Buffalo, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Stony Brook University, Stony Brook, New York
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Mayfield Clinic, Cincinnati, Ohio
  - Ohio State University, Columbus, Ohio
  - Medical Center of South Carolina, Charleston, South Carolina
  - Prisma Health, Greenville, South Carolina
  - Tennessee Interventional Associates - Erlanger, Chattanooga, Tennessee
  - Fort Sanders Regional Medical Center, Knoxville, Tennessee
  - University of Tennessee Medical Center - Knoxville, Knoxville, Tennessee
  - Methodist University Hospital, Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas - Southwestern, Dallas, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - West Virginia University Hospital, Morgantown, West Virginia

REFERENCES:
- See also: Vanderbilt University Medical Center-Department of Neurological Surgery — https://www.vumc.org/neurosurgerydept/welcome

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT01655784/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/84/NCT01655784/ICF_001.pdf